CLINICAL TRIAL: NCT06588023
Title: Prevalence of Blood Pressure Complications During Cesarean Section in Pre-eclamptic Patients
Brief Title: Prevalence of Blood Pressure Complications During Cesarean Section in Pre-eclamptic Patients (HOPE)
Acronym: HOPE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: M24BM0715
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pre-eclampsia; Pre-Eclampsia, Severe
Keywords: cesarean section; Blood pressure complications; pre-eclampsia; hypertension; hypotension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lille University Hospital: Pre-eclamptic patients undergoing a cesarean section at the maternity ward of Lille University Hospital.
  Interventions: Other: Observational study to evaluate professional practices
- Clermont-Ferrand University Hospital: Pre-eclamptic patients undergoing a cesarean section at the maternity ward of Clermont-Ferrand University Hospital.
  Interventions: Other: Observational study to evaluate professional practices

INTERVENTIONS:
Other: Observational study to evaluate professional practices — It consists of collecting data prospectively on all pre-eclamptic patients undergoing a non-urgent cesarean section.
  The objective is to observe the management of hemodynamics and calculate the prevalence of complications such as maternal hypotension and/or hypertension through the implementation of non-invasive monitoring (ClearSight).

SUMMARY:
Preeclampsia (PE) is an obstetric placental vascular pathology with a prevalence of 2 to 5% of pregnant women. It is defined by learned societies by the association of high blood pressure (BP≥140/90mmHg) and proteinuria > 0.3g/day. The last French Maternal Mortality Report 2024 places cardiovascular complications among the main causes of maternal death. PE has an increasing number of deaths in 2016-2018 and significant preventability (66%).

Cesarean sections in pre-eclamptic patients are difficult procedures and, do not benefit from any specific recommendations. Cesarean section is promptly performed under regional anesthesia by spinal anesthesia or spinal anesthesia with combined epidural, techniques that cause maternal arterial hypotension with consequences for the baby.

These hypertensive patients, often on antihypertensives, challenge the anesthesiologist to manage the hemodynamic balance between the risk of arterial hypotension generated by the anesthesia corrected by vasoactive amines and the risk of major hypertension secondary to their management. The major risk in these patients with low platelet counts is hemorrhagic stroke.

Our study is an observational, bi-centric study between the maternity wards of the Clermont Ferrand and Lille University Hospitals.

It consists of collecting data prospectively on all pre-eclamptic patients undergoing a non-urgent cesarean section.

The objective is to observe the management of hemodynamics and calculate the prevalence of complications such as maternal hypotension and/or hypertension through the implementation of non-invasive monitoring (ClearSight).

Patients meeting the inclusion and non-inclusion criteria may be included in the study by an investigator after having given a non-opposition agreement after having received clear and fair information about the study.

In any case, the care of patients participating in the study will not be modified in any way compared to the usual practices of the services.

ELIGIBILITY:
Inclusion Criteria:

* Pre-eclamptic patient according to the criteria defined by SFAR 2020.
* Indication of organised or semi-urgent cesarean section (Green or Orange code).
* Adult patient, benefiting from a social security system.
* Oral non-opposition to participation in the study.

Exclusion Criteria:

* Urgent Cesarean (Red code).
* Patient refusal.
* Patient does not understand French.
* Individual protection measures : guardianship, curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-eclamptic patients undergoing cesarean section in the maternity wards of the Clermont-Ferrand and Lille university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic events. | During the entire cesarean procedure including anesthesia.
  Prevalence of the occurrence of events such as maternal arterial hypotension and/or arterial hypertension during a cesarean section in a known pre-eclamptic patient.

SECONDARY OUTCOMES:
Duration of maternal hypotensive or hypertensive episodes. | During the entire cesarean procedure including anesthesia.
  Defined by the time-weighted average intraoperative PAS below a threshold of 110mmHg or above a threshold of 170mmHg. This measurement is commonly called TWA (Time Weighted Average), corresponding to the area between the chosen PAS threshold and the measured PAS curve, divided by the total measurement time.
Number of maternal hypotensive and/or hypertensive episodes. | During the entire cesarean procedure including anesthesia.
Occurrence of major adverse events. | During the entire cesarean procedure including anesthesia.
Nature and dose of local anesthetic administered | During the entire cesarean procedure including anesthesia.
Nature and management of antihypertensive drugs during cesarean section. | During the entire cesarean procedure including anesthesia.

OTHER OUTCOMES:
Maximum dosages and cumulative doses of Noradrenaline during cesarean section. | During the entire cesarean procedure including anesthesia.
Total vascular filling volume. | During the entire cesarean procedure including anesthesia.
Total diuresis. | During the entire cesarean procedure including anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: MARTINE BONNIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided